CLINICAL TRIAL: NCT06794203
Title: Hyperthyroidism in the Immediate Post-kidney Transplantation Period: a Potential Predictive of Worse Outcome of Renal Graft
Brief Title: Hyperthyroidism as a Potential Predictive of Worse Outcome of Renal Graft
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ITTX-21
Record Dates: First submitted 2024-12-30; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Kidney Diseases; Kidney Transplant; Hyperthyroidism
Keywords: Hyperthyroidism; Kidney Diseases
MeSH Terms: conditions — Kidney Diseases; Hyperthyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney transplant patients: All kidney transplant patients at the U.O. of Nephrology, Dialysis and Transplantation directed by Prof. Gaetano La Manna of the Policlinico Sant'Orsola - IRCCS Azienda Ospedaliero Universitaria of Bologna.

SUMMARY:
The objectives of the study are: to research the association, if any, between the occurrence of thyroid function changes in the immediate post-transplant period and the prognosis of the transplant itself; identify any risk factors for the occurrence of thyroid disorders In the immediate post-transplant period.

DETAILED DESCRIPTION:
Kidney transplant patients are by definition affected by MRC, regardless of eGFR. However, at the same time, several factors make them a unique category with distant characteristics from non-kidney transplant MRC patients.

Immunosuppressant and corticosteroid therapy could affect a variety of systems, including the pituitary-thyroid-kidney axis. MTOR inhibitors, for example, would result in increased iodine uptake in TSH-stimulated thyrocytes.

Corticosteroids, on the other hand, inhibit the conversion of T4 to T3 and inhibit the TSH production in a dose-dependent manner, and this activity could contribute to the low T3 syndrome that some sturi repot in the phase immediately following kidney transplantation.

In addition, abrupt changes in the serum concentration of thyroid hormones in the immediate post kidney transplantation could be influenced by the stress surgery related to the surgery itself and by exposure to iodinated agents (antiseptics and iodinated contrast medium).

The objectives of the study are:

1. To research the association, if any, between the occurrence of thyroid function changes in the immediate post-transplant period and the prognosis of the transplant itself in terms of:

   * Renal function three months after transplantation.
   * Medical complications in the post-transplant period (from surgery to patient discharge)
   * Patient survival at three months after transplantation.
2. Identify any risk factors for the occurrence of thyroid disorders In the immediate post-transplant period.

During the past 5 years at the Transplant Center of the Nephrology OU, Dialysis, Transplantation of our hospital, 579 kidney transplants have been performed with an average of about 115 transplants per year. It is therefore estimated for our study a sample size of about 100 patients, given the need to meet the inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects transplanted at our Center;
* Subjects whose 3-month follow-up is available;
* Age ≥18 years;
* Availability of clinical and laboratory data regarding thyroid function trends in the immediate post-transplant period (within 30 days after transplantation);
* Subjects giving informed consent to participate.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All kidney transplant patients at the U.O. of Nephrology, Dialysis and Transplantation directed by Prof. Gaetano La Manna of Policlinico Sant'Orsola - IRCCS Azienda Ospedaliero Universitaria di Bologna.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Thyroid function | At baseline, then 3-month follow-up after kidney transplantation
  To research, if any, the alteration of thyroid function in the immediate post-transplant period
Renal function | At 3-month follow-up after kidney transplantation
  Investigating renal function three months after transplantation.
Medical complications | Baseline (surgery), at 3-month follow-up after kidney transplantation, at patient discharge
  Investigate about medical complications in the post-transplant period
Survival | At 3-month follow-up after kidney transplantation
  Patient survival at three months after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano La Manna, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, BO, Italy